CLINICAL TRIAL: NCT01023230
Title: A Phase Ib Dose-Escalation Study to Assess the Safety and Tolerability of DV-601 in Subjects With Chronic Hepatitis B on Concurrent Treatment With a Nucleoside Analogue
Brief Title: A Study to Assess DV-601 in Subjects With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DV4-HBT-02; 2009-010142-66 (Registry Identifier: EudraCT)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Hepatitis B, Chronic
Keywords: DV-601; hepatitis B; entecavir; therapeutic vaccine
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DV-601 (Experimental)
  Interventions: Drug: DV-601; Drug: Entecavir

INTERVENTIONS:
Drug: DV-601 — Six injections of DV-601 administered over a period of 12 weeks.
Drug: Entecavir — Daily dosing starting approximately 4 weeks prior to first dose of DV-601 for one year total duration.
  Other Names: Baraclude

SUMMARY:
The purpose of this study is to determine if DV-601, an investigational, therapeutic vaccine will be well-tolerated and induce hepatitis B virus (HBV)-specific virological and immunological responses in chronic hepatitis B (CHB) patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 to 65 years of age.
* Signed informed consent.
* Diagnosis of CHB and candidates for therapy
* Normal renal function
* Women of childbearing potential must have a serum negative pregnancy test at screening. Women of childbearing potential and males whose sexual partners are of childbearing potential must agree to use dual methods of contraception.

Exclusion Criteria:

* Liver disease other than CHB
* Documented co-infection with hepatitis A virus (HAV), hepatitis C virus (HCV), or HIV
* Previous therapy with interferon alpha.
* Any other antiviral therapy for chronic hepatitis B within the previous 3 months prior to Screening Visit.
* Immunosuppressive treatment (e.g. chemotherapy, high-dose of steroids) within 6 months of Screening Visit.
* Evidence of cirrhosis
* Child-Turcotte-Pugh (CTP) score ≥ 7, either currently or at any occasion in the past
* Clinically significant acute or chronic illnesses, such as autoimmune diseases, collagen vascular disease, immune deficiencies, active or uncontrolled infections, etc. as determined by the investigator and documented in medical history.
* Malignancy other than curatively treated, superficial skin cancer or carcinoma in situ of the cervix.
* Participation in any experimental protocol or therapy within 28 days prior to the Screening Visit.
* Current substance or alcohol abuse that in the opinion of the investigator would interfere with compliance or with interpretation of study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Patient diaries, adverse events, physical exams, and lab tests | Through Day 99

SECONDARY OUTCOMES:
HBV-DNA levels | Change from baseline to Days 43 and 99, and to Weeks 24 and 48

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (4):
  - Collegium Medicum Uniwersytet im. Mikołaja Kopernika, Bydgoszcz
  - Samodzielny Publiczny Wojewódzki Szpital Zespolony, Szczecin
  - Wojewódzki Szpital Zakaźny, Warsaw
  - NZOZ Centrum Badan Klinicznych, Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided
a/o August 2016, decision is still pending.